CLINICAL TRIAL: NCT04494113
Title: A Phase 0 Window-of-Opportunity Pharmacodynamic Trial of Triapine (NSC# 663249) in Uterine Corpus Serous Adenocarcinoma
Brief Title: Testing the Response to the Anti-cancer Drug, Triapine, in Uterine Cancers Using Markers From the Tissue at the Time of Hysterectomy
Status: Suspended | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Other - evaluation of enrolled patients
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-05457; NCI-2020-05457 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10401 (Other: JHU Sidney Kimmel Comprehensive Cancer Center LAO); 10401 (Other: CTEP); UM1CA186691 (NIH)
Record Dates: First submitted 2020-07-30; First posted 2020-07-31 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Endometrial Serous Adenocarcinoma
MeSH Terms: interventions — Biopsy; Specimen Handling; 3-aminopyridine-2-carboxaldehyde thiosemicarbazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (triapine, surgical resection) (Experimental): Patients receive triapine IV over 2 hours on day 1. Patients then undergo surgical resection and tissue collection 6-8 hours after the initiation of the triapine infusion. Patients also undergo biopsy and collection of blood samples on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Resection; Drug: Triapine

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of tissue and blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Resection — Undergo surgical resection
  Other Names: Surgical Resection
Drug: Triapine — Given IV
  Other Names: 3-aminopyridine-2-carboxaldehyde thiosemicarbazone; 3-AP; 3-Apct; OCX-0191; OCX-191; OCX191; PAN-811

SUMMARY:
This early phase I trial investigates the response to the anti-cancer drug, triapine, in uterine cancers by using markers from tissue samples at the time of removal of the uterus, ovaries, and fallopian tubes (hysterectomy and bilateral salpingo-oophorectomy). Triapine may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Adding triapine to the usual approach of surgery followed by chemotherapy alone or in combination with radiation therapy may help to slow the growth of uterine cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine whether intravenous (IV) triapine 25 mg/m^2 will induce cell cycle arrest as measured by phospho-histone H3 (pHH3) in uterine serous adenocarcinoma cells removed at the time of hysterectomy.

SECONDARY OBJECTIVES:

I. Determine whether a preoperative dose of intravenous triapine 25 mg/m^2 can be safely given prior to hysterectomy and staging for uterine serous adenocarcinoma.

II. Determine whether changes in cyclin D/E and Ki-67 protein expression are detectable using immunohistochemistry pre- and post-triapine treatment in uterine serous adenocarcinomas.

III. Evaluate plasma and tissue triapine concentrations.

EXPLORATORY OBJECTIVES:

I. Determine the feasibility of using single-cell transcriptome analysis to quantify changes in gene expression following triapine treatment and to evaluate their concordance with immunohistochemistry (IHC) endpoints of cell cycle arrest.

II. Identify genomic variants of uterine serous adenocarcinoma (including but not limited to p53) with treatment response to ribonucleotide reductase inhibitors such as triapine using whole exome sequencing (WES).

OUTLINE:

Patients receive triapine IV over 2 hours on day 1. Patients then undergo surgical resection and tissue collection 6-8 hours after the initiation of the triapine infusion. Patients also undergo biopsy and collection of blood samples on study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed uterine corpus serous adenocarcinoma
* Patients must be planned for surgical hysterectomy and operative staging
* Patients must have adequate archival tissue obtained within 8 weeks of step 1 registration OR have sufficient tumor tissue and be willing to undergo an endometrial pipelle biopsy prior to beginning study treatment.
* Patients must have adequate primary tumor volume, as determined by imaging (e.g., computed tomography [CT], ultrasound, magnetic resonance imaging [MRI]) at eligibility screening, to accommodate research specimen collections in addition to clinical pathology evaluation
* Patients must not have received any prior anticancer treatment for endometrial cancer
* Patients must be >= 18 years old. Because no dosing or adverse event data are currently available on the use of triapine in patients < 18 years of age, children are excluded from this study
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Absolute neutrophil count >= 1,000/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9.0 g/dL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional ULN
* International normalized ratio (INR) =< 2
* Creatinine =< 1.5 x institutional ULN OR glomerular filtration rate (GFR) >= 60 mL/min/1.73 m^2 unless data exists supporting safe use at lower kidney function values, no lower than 30 mL/min/1.73 m^2
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Patients of childbearing potential must have a negative pregnancy test result prior to beginning study treatment
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity (IDMC) are not eligible as there is limited likelihood of direct benefit for participants in this study

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia
* Patients who are receiving any other investigational agents
* Patients who have known brain metastases, as they are not candidates for surgery
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to triapine
* Patients receiving any medications or substances that are inhibitors or inducers of triapine, as well as medications known to be associated with methemoglobinemia, are ineligible. Triapine drug interactions have not yet been identified. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Patients with uncontrolled intercurrent illness
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Patients with glucose-6-phosphate dehydrogenase (G6PD) deficiency are not eligible. Patients at risk for G6PD deficiency must be screened prior to enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-02-08 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Pharmacodynamic response | Up to 6-8 hours post-triapine infusion
  Pharmacodynamic response rate will be estimated as the proportion of evaluable patients who achieve pharmacodynamic response defined as a decrease in phospho-histone H3 immunoscore of >= 1 from baseline to post-exposure of intravenous triapine for each patient. The corresponding 95% confidence interval will be provided.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to day 42
  Dose-limiting toxicities, as listed by Common Terminology Criteria for Adverse Events, version 5, are defined as any pre-surgical grade 3 or higher non-hematologic toxicity or grade 4 neutropenia, neutropenic fever, or thrombocytopenia within 24 hours of triapine administration. Toxicity will be tabulated by type and grade.
Pharmacokinetic (PK) analysis | Baseline, 5 minutes before end of triapine infusion, 6-8 hours post-infusion (at time of surgical tissue resection), and 24 hours post-infusion
  End of infusion plasma concentrations represent maximum concentration and will be compared with historical data. Post-triapine plasma and tissue concentrations will generate plasma to tissue ratios, which represent the tissue partitioning coefficient, a useful PK parameter.

OTHER OUTCOMES:
Single-cell transcriptome analysis | Baseline, post-triapine infusion, surgical resection
  Single-cell transcriptome analysis will be conducted to quantify changes in gene expression following triapine treatment. Changes of gene expression will be correlated with immunohistochemistry endpoints of cell cycle arrest.
Whole exome sequencing (WES) analysis | Baseline
  WES will be used to identify genomic variants of uterine serous adenocarcinoma (including but not limited to p53) that can predict the treatment response to triapine.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca L Stone, Principal Investigator — JHU Sidney Kimmel Comprehensive Cancer Center LAO
Locations (7):
- United States (7):
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm